CLINICAL TRIAL: NCT05513001
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized Withdrawal and Open-label Extension Study Followed by Long-term Open-label Treatment Cycles to Assess the Efficacy, Safety and Tolerability of Remibrutinib (LOU064) in Adult Chronic Spontaneous Urticaria Patients Who Completed the Preceding Remibrutinib Phase 3 Studies
Brief Title: An Extension Study of Long-term Efficacy, Safety and Tolerability of Remibrutinib in Chronic Spontaneous Urticaria Patients Who Completed Preceding Studies With Remibrutinib
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLOU064A2303B; 2022-001034-11 (EudraCT Number)
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: CSU; Brutons Tyrosine Kinase (BTK) inhibitor; Chronic Spontaneous Urticaria; Urticaria activity score; Hives severity score; Itch severity score; Extension; Randomized withdrawal; Retreatment upon relapse; Remibrutinib
MeSH Terms: conditions — Chronic Urticaria | interventions — remibrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: LOU064 (blinded) (Experimental): LOU064 (blinded) taken orally for 24 weeks, followed by cycles of either LOU064 (open-label) taken orally for a maximum of 5 cycles of 24 weeks each OR treatment-free observation cycles. Randomized in a 1:1 ratio (arm 1:arm 2)
  Interventions: Drug: LOU064 (blinded); Drug: LOU064 (open label)
- Arm 2: LOU064 Placebo (blinded) (Placebo Comparator): LOU064 placebo (blinded) taken orally for 24 weeks, followed by cycles of either LOU064 (open-label) taken orally for a maximum of 5 cycles of 24 weeks each OR treatment-free observation cycles. Randomized in a 1:1 ratio (arm 1:arm 2)
  Interventions: Drug: Placebo; Drug: LOU064 (open label)
- Arm 3: LOU064 (Open Label) (Experimental): LOU064 (open-label) taken orally for 24 weeks per treatment cycle (Arm 3)
  Interventions: Drug: LOU064 (open label)

INTERVENTIONS:
Drug: LOU064 (blinded) — LOU064 (blinded) active treatment
  Other Names: remibrutinib
  Arms: Arm 1: LOU064 (blinded)
Drug: Placebo — Placebo
  Arms: Arm 2: LOU064 Placebo (blinded)
Drug: LOU064 (open label) — LOU064 (open-label) active treatment
  Other Names: remibrutinib

SUMMARY:
The purpose of this extension study is to collect long-term efficacy, safety and tolerability data on remibrutinib in a selected group of participants with Chronic Spontaneous Urticaria (CSU) who previously completed the treatment phase of remibrutinib preceding Phase 3 core studies.

This study will also fulfill the Novartis commitment to provide post-trial access to participants who have completed the preceding Phase 3 studies, where applicable.

DETAILED DESCRIPTION:
This is a Phase 3b multicenter, double-blind, placebo-controlled, randomized withdrawal, and open-label extension study to evaluate the efficacy and safety of remibrutinib 25 mg twice daily (b.i.d.) in adult CSU participants who have completed one of the preceding Phase 3 core studies. The study comprises 2 Epochs:

Epoch 1 is the initial study period and includes participants from preceding Phase 3 studies. It consists of a 24-week randomized withdrawal period where participants receive either remibrutinib 25 mg b.i.d. or placebo if their UAS7 score is less than 16. For those with a UAS7 score of 16 or higher, there is a 24-week open-label treatment period with remibrutinib 25 mg b.i.d. Participants are randomized 1:1 to the double-blind placebo-controlled withdrawal phase. All participants will continue their background H1-AH treatment. If participants relapse (UAS7 ≥ 16) in the blinded group, they enter the (Re-)treatment period of Epoch 1 and receive 24 weeks of open-label treatment with remibrutinib 25 mg b.i.d. After this period, they move to Epoch 2.

Epoch 2 is the second subsequent study period and consists of 24-week cycles that may include treatment-free observation and/or open-label (Re-)treatment periods with remibrutinib 25 mg b.i.d., with or without background H1-AH, at the investigator's discretion. Participants from future Phase 3 remibrutinib studies may also join Epoch 2 if approved. If participants relapse (UAS7 ≥ 16) during an observation period, they enter the next (Re-)treatment period for 24 weeks of treatment with remibrutinib 25 mg b.i.d. Participants completing an observation period with a UAS7 ≤ 6 will complete the study with an end-of-study (EOS) visit. Those with a UAS7 > 6 but < 16 can enter the next (Re-)treatment period if continuous treatment is deemed necessary. Participants with a UAS7 < 16 in the previous treatment period will receive remibrutinib monotherapy (without background H1-AH). If treatment continuation is not necessary, they complete the EOS visit and leave the study. Participants with a UAS7 ≥ 16 during the observation period will enter the corresponding (Re-)treatment period to continue treatment.

Throughout Epoch 2, the use of background H1-AH is at the investigator's discretion, except for participants with a UAS7 < 16 in the previous treatment period, who will be treated with remibrutinib monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Male and female, adult participants ≥18 years of age.
* Participants who successfully completed the preceding core studies CLOU064A2301, CLOU064A2302, CLOU064A1301, CLOU064A2304 or CLOU064A2305 according to the respective protocols.
* Willing and able to adhere to the study protocol and visit schedule.

Exclusion Criteria:

* Significant bleeding risk or coagulation disorders.
* History of gastrointestinal bleeding.
* Requirement for anti-platelet medication.
* Requirement for anticoagulant medication.
* History or current hepatic disease.
* Evidence of clinically significant cardiovascular, neurological, psychiatric, pulmonary, renal, hepatic, endocrine, metabolic, hematological disorders, gastrointestinal disease or immunodeficiency that, in the investigator's opinion, would compromise the safety of the participant, interfere with the interpretation of the study results or otherwise preclude participation or protocol adherence of the participant.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2027-08-02 (Estimated)

PRIMARY OUTCOMES:
Time to first composite event (i.e., relapse (UAS7≥16) | 24 weeks
  The efficacy of remibrutinib in CSU participants with a UAS7<16 at Week 52 in the prior core study with respect to time to first of the three events: relapse or study treatment discontinuation due to lack of efficacy or intake of strongly confounding prohibited medication up to Week 24 compared to placebo. (Epoch 1)
  Time to first composite event (i.e., relapse (UAS7≥16), study treatment discontinuation due to lack of efficacy or intake of strongly confounding prohibited medication) during the randomized withdrawal period (Epoch 1)
  Urticaria Activity Score (UAS7) describes the number of hives with 0 being No Hives and 3 is most severe. The final score is calculated by adding together daily scores which can range from 0-6 for 7 days. The resulting maximum score is then 42.

SECONDARY OUTCOMES:
Number of participants with treatment-emergent (serious and non-serious) adverse events | 160 weeks
  Occurrence of treatment-emergent (serious and non-serious) adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (179):
- United States (43):
  - Allervie Clinical Research, Birmingham, Alabama
  - Cahaba Derm and skin hlth ctr 27, Birmingham, Alabama
  - Research Solutions of Arizona, Litchfield Park, Arizona
  - Acuro Research Inc, Little Rock, Arkansas
  - Arkansas Research Trials, North Little Rock, Arkansas
  - Kern Research, Bakersfield, California
  - Antelope Valley Clinical Trials, Lancaster, California
  - Allergy and Asthma Consultants, Redwood City, California
  - Asthma and Allergy Associates P C, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Ctr PC, Denver, Colorado
  - UCONN Health Dermatology, Farmington, Connecticut
  - Florida Ctr Allergy Asthma Research, Aventura, Florida
  - Finlay Medical Research, Greenacres City, Florida
  - Miami Dade Medical Research, Miami, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - Allergy and Asthma Diagnostic Treatment Center, Tallahassee, Florida
  - AeroAllergy Research Laboratories of Savannah Inc, Savannah, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Endeavor Health, Glenview, Illinois
  - Asthma and Allergy Center of Chicago S C, River Forest, Illinois
  - Deaconess Clin Allerg Res Inst, Evansville, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Allergy and Asthma Specialist P S C, Owensboro, Kentucky
  - John Hopkins University, Baltimore, Maryland
  - Institute for Asthma and Allergy PC, Chevy Chase, Maryland
  - The Clinical Research Center, St Louis, Missouri
  - Somnos Clinical Research, Lincoln, Nebraska
  - Allergy Asthma Assoc Monmouth, Little Silver, New Jersey
  - Oakview Dermatology, Athens, Ohio
  - Optimed Research LLC, Columbus, Ohio
  - CR Services Acquisition US, Dublin, Ohio
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - Allergy Asthma and Clinical Research, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, Tulsa, Oklahoma
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - National Allergy and Asthma Research LLS, North Charleston, South Carolina
  - Orion Clinical Research, Austin, Texas
  - Western Sky Medical Research, El Paso, Texas
  - RFSA Dermatology, San Antonio, Texas
  - Allergy Associates of Utah, Sandy City, Utah
  - Bellingham Asthma Allergy and Immunology, Bellingham, Washington
  - Seattle Allergy and Asthma Rsch, Seattle, Washington
  - Allergy Asthma and amp Sinus Ctr S C, Greenfield, Wisconsin
- Argentina (7):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Buenos Aires, Nueve De Julio
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Bahía Blanca
  - Novartis Investigative Site, Capital Federal
  - Novartis Investigative Site, Santa Fe
- Australia (2):
  - Novartis Investigative Site, East Melbourne, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Novartis Investigative Site, Santo André, São Paulo, Brazil
- Bulgaria (2):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
- Canada (9):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Fredericton, New Brunswick
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Niagara Falls, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Verdun, Quebec
- China (10):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Guangdong, Guangzhou
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Wuxi, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Colombia (3):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bogotá
- Czechia (4):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Plzen Bory
  - Novartis Investigative Site, Prague
- Denmark (2):
  - Novartis Investigative Site, Hellerup
  - Novartis Investigative Site, Kobenhavn N V
- France (12):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Antony
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Mandé
  - Novartis Investigative Site, Toulouse
- Germany (13):
  - Novartis Investigative Site, Bramsche, Lower Saxony
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Merzig, Saarland
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
- Hungary (2):
  - Novartis Investigative Site, Debrecen, Hajdú-Bihar
  - Novartis Investigative Site, Debrecen
- Novartis Investigative Site, Belagavi, Karnataka, India
- Italy (2):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Milan, MI
- Japan (16):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Urayasu, Chiba
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kamimashi-gun, Kumamoto
  - Novartis Investigative Site, Izumiōtsu, Osaka
  - Novartis Investigative Site, Neyagawa, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Koto, Tokyo
  - Novartis Investigative Site, Minato, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Osaka
- Malaysia (5):
  - Novartis Investigative Site, Muar town, Johor
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Ipoh, Perak
  - Novartis Investigative Site, George Town, Pulau Pinang
  - Novartis Investigative Site, Wilayah Persekutuan
- Poland (4):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- Alma Cruz-Santana Private Practice, Carolina, Puerto Rico
- Russia (4):
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Stavropol
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (6):
  - Novartis Investigative Site, Kežmarok
  - Novartis Investigative Site, Komárno
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Svidník
- South Africa (2):
  - Novartis Investigative Site, Pretoria, Gauteng
  - Novartis Investigative Site, Cape Town, Western Province
- South Korea (6):
  - Novartis Investigative Site, Daegu, Dalseo Gu
  - Novartis Investigative Site, Hwaseong-si, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Zurich
- Taiwan (3):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Thailand (3):
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (7):
  - Novartis Investigative Site, Aydin
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kayseri
  - Novartis Investigative Site, Sakarya
  - Novartis Investigative Site, Samsun
  - Novartis Investigative Site, Talas Kayseri
- Novartis Investigative Site, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com